CLINICAL TRIAL: NCT01094860
Title: A Pharmacokinetic and Pharmacodynamic Study to Evaluate the Safety and Feasibility of Continuous Infusion Nelarabine in Patients With Relapsed / Refractory Lymphoid Malignancies
Brief Title: Pharmacokinetic (PK) and Pharmacodynamic (PD) Study of Nelarabine in Patients With Relapsed/Refractory Lymphoid Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2009-0717; NCI-2010-01659 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2010-03-25; First posted 2010-03-29 (Estimated); Last update posted 2020-02-11 (Actual); Status verified 2020-02

CONDITIONS: Leukemia
Keywords: Relapsed/Refractory Lymphoid Malignancies; Chronic lymphocytic leukemia; CLL; Small lymphocytic lymphoma; SLL; B-prolymphocytic leukemia; Follicular lymphoma; Mantle cell lymphoma; Lymphoplasmacytoid lymphoma; Marginal zone lymphoma; T-cell prolymphocytic leukemia; large granular lymphocyte leukemia; mycosis fungoides; Sezary syndrome; peripheral T-cell lymphoma; Chemotherapy; Monoclonal antibody therapy; T-cell or B-cell acute lymphoblastic leukemia (ALL); Continuous Infusion Nelarabine; Arranon
MeSH Terms: conditions — Leukemia; Recurrence; Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia, Prolymphocytic, B-Cell; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Waldenstrom Macroglobulinemia; Lymphoma, B-Cell, Marginal Zone; Leukemia, Prolymphocytic, T-Cell; Leukemia, Large Granular Lymphocytic; Mycosis Fungoides; Sezary Syndrome; Lymphoma, T-Cell, Peripheral; Leukemia, Biphenotypic, Acute | interventions — nelarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Continuous Infusion Nelarabine (Experimental): Starting dose 200 mg/m2 x 5 days
  Interventions: Drug: Nelarabine

INTERVENTIONS:
Drug: Nelarabine — Starting dose 200 mg/m2 for 5 day continuous infusion administered via a central catheter, repeated every 28 days.
  Other Names: Arranon

SUMMARY:
The goal of the clinical research study is to find the highest tolerable dose of nelarabine when given as a continuous infusion to patients with a lymphoid malignancy that has not responded to, or has come back after treatment with chemotherapy. The safety of this drug will also be studied.

DETAILED DESCRIPTION:
The Study Drug:

Nelarabine is designed to interfere with DNA (the genetic material of cells) and stop the growth of rapidly dividing cells, such as cancer cells.

Study Groups:

If you are found to be eligible to take part in this study, you will be assigned to a dose level of nelarabine based on when you joined this study. Up to 8 dose levels of nelarabine will be tested. Three (3) to 6 participants will be enrolled at each dose level. The first group of participants will receive the lowest dose level. Each new group will receive a higher dose than the group before it, if no intolerable side effects were seen. This will continue until the highest tolerable dose of nelarabine is found.

Study Drug Administration:

You will receive nelarabine as a non-stop infusion through a needle or catheter in your vein on Days 1-5 of each 4 - 6 week cycle. You will remain in the hospital for this infusion.

You may receive ondansetron or a similar drug by vein over about 30 minutes before you receive nelarabine. This is given to help prevent nausea. You will also take ondansetron or a similar drug by mouth every 12 hours for the next 7 days as needed. If you are still having nausea, you will be given additional drugs.

If you are not allergic, you may receive allopurinol by mouth on Days 1-10 of Cycles 1. Allopurinol is given to help reduce the risk of too much uric acid in the blood. If the level of uric acid in the blood is too high, you may receive additional drugs.

You may also be given drugs to help reduce the risk of infection.

Study Visits:

On Day 1 of Cycle 1 only, blood (about 2 teaspoons each time) will be drawn for pharmacokinetic (PK) and pharmacodynamic (PD) testing 1 hour before, then again 2, 4, 6, and between 10-18 hours after the study drug infusion. PK testing measures the amount of study drug in the body at different time points. PD testing measures how the level of study drug in your body may affect the disease

On Days 2, 3, 4, and 5 of Cycle 1 only, blood (about 2 teaspoons) will be drawn for PK and PD testing.

On Day 1 of each cycle:

* You will have a physical exam, including measurement of your vital signs.
* You will be asked about any drugs you are taking and about any transfusions you may have had.
* You will be asked about any side effects you may have had.
* Your performance status will be recorded.
* Measurements of your lymph nodes, spleen, and liver will be taken.
* Blood (about 2 teaspoons) will be drawn to test the levels of antibodies and T-cells (a type of white blood cell) in your blood.

One (1) time each week, or more often if the study doctor thinks it is needed:

* You will have a physical exam, including measurement of your vital signs.
* You will be asked about any side effects you may have had.
* Your performance status will be recorded.
* Blood (about 4 teaspoons) will be drawn for routine tests.

After every 3 cycles:

* You will have a physical exam, including measurement of your vital signs.
* You will be asked about any drugs you are taking and about any transfusions you may have had.
* You will be asked about any side effects you may have had.
* Your performance status will be recorded.
* Measurements of your lymph nodes, spleen, and liver will be taken.
* Blood (about 4 teaspoons) will be drawn for routine tests.
* You will have a neurological exam (tests to check the functioning of your nerves, including tests of your balance and reflexes).
* Blood (about 2 teaspoons) will be drawn to check the number of T-cells in your blood.
* You will have a bone marrow aspirate/biopsy to check the status of the disease.
* If you have NHL, you will have CT scan of the chest, abdomen, and pelvis to check the status of the disease.

Length of Participation:

You may continue to receive nelarabine for as long as the study doctor thinks it is in your best interest. You will no longer be able to receive the study drug if the disease gets worse or intolerable side effects occur.

This is an investigational study. Nelarabine, given as an injection, is FDA approved for the treatment of refractory or relapsed T-cell acute lymphoblastic leukemia or T lymphoblastic lymphoma. The use of nelarabine as a continuous infusion is investigational.

Up to 35 patients will take part in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have one of the following relapsed/ refractory lymphoid malignancies: Chronic lymphocytic leukemia (CLL), small lymphocytic lymphoma (SLL) or B-prolymphocytic leukemia which has been previously treated with a purine analog, and are not candidates for higher priority clinical studies. Follicular lymphoma, mantle cell lymphoma, lymphoplasmacytoid lymphoma or marginal zone lymphoma which has been previously treated with autologous or allogeneic stem cell transplantation.
2. Continued from #1:T-cell prolymphocytic leukemia, large granular lymphocyte leukemia, mycosis fungoides / Sezary syndrome or peripheral T-cell lymphoma which has been previously treated with at least one line of chemotherapy or monoclonal antibody therapy. T-cell or B-cell acute lymphoblastic leukemia (ALL) which has been previously treated with at least one line of chemotherapy.
3. Patients (both pediatrics and adults) must have adequate renal function (calculated creatinine clearance >/= 50ml/min). For adults this will be calculated per the Cockcroft -Gault formula and in pediatric cases this will be calculated per the Schwartz formula.
4. Patients must have adequate hepatic function (bilirubin </= 2 mg/dL; SGOT or SGPT </= 3X the ULN for the reference lab unless due to leukemia).
5. Patients must have adequate marrow function (neutrophils >/= 0.5x10^9/L and platelets >/= 50x10^9/L) unless cytopenias are deemed due to disease.
6. Patients must have adequate performance status (Zubrod 0-2).
7. Female patients must not be pregnant or lactating. Female patients of childbearing potential (including those <1 year postmenopausal) and male patients must agree to use contraception.
8. Patients must sign an informed consent form indicating that they are aware of the investigational nature of this study, in keeping with the policies of the hospital.

Exclusion Criteria:

1. Patients must not have untreated or uncontrolled life-threatening infection.
2. Patients known to be HIV positive or known to have Hepatitis B and/or C are excluded.
3. Patients must not have received systemic chemotherapy or monoclonal antibody therapy within 2 weeks of study enrollment. Patients who have previously received bolus nelarabine are still eligible. Hydroxyurea or corticosteroids for control of blood counts is allowed, but must be discontinued 24 hours prior to initiating nelarabine.
4. Patients must not have a history of grade >/=2 neurological toxicity with previous treatment, or persistent grade >/=2 peripheral neuropathy. Drowsiness and lethargy were exempted from this criteria unless previously persistent for more than one week.
5. Patients must not have uncontrolled central nervous system disease. Patients with a history of seizure disorders must be seizure-free for one year prior to enrolment.
6. Patients must not have any other medical condition, including mental illness or substance abuse, deemed by the Investigator to be likely to interfere with a patient's ability to give informed consent or cooperate and participate in the study or interfere with the interpretation of the results.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2010-06-08 (Actual); Primary Completion 2018-08-09 (Actual); Study Completion 2018-08-09 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) of a 5-day Continuous Infusion Schedule of Nelarabine | 28 day cycle
  MTD defined as the highest dose that no more than 1 dose limiting toxicity (DLT) occurs among 6 patients. Dose-limiting toxicity (DLT) defined based on drug related events only. DLT in the first treatment cycle used for the dose escalation.

CONTACTS AND LOCATIONS:
Overall Officials: Tapan Kadia, MD, Study Chair — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Boddu PC, Senapati J, Ravandi-Kashani F, Jabbour EJ, Jain N, Ayres M, Chen Y, Keating MJ, Kantarjian HM, Gandhi V, Kadia TM. A phase 1 study to evaluate the safety, pharmacology, and feasibility of continuous infusion nelarabine in patients with relapsed and/or refractory lymphoid malignancies. Cancer. 2023 Feb 15;129(4):580-589. doi: 10.1002/cncr.34570. Epub 2022 Nov 29. PMID 36448227
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org